CLINICAL TRIAL: NCT01185743
Title: Effect of Atypical Antipsychotics on Gene Expression in Soft Tissues of Healthy Subjects - A Placebo Controlled Randomised Pilot Study
Brief Title: Antipsychotics and Gene Expression in Soft Tissues
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Martin Bauer, MD, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: OLA_ZIPRA
Record Dates: First submitted 2010-08-19; First posted 2010-08-20 (Estimated); Last update posted 2017-03-23 (Actual); Status verified 2017-03

CONDITIONS: Schizophrenia; Diabetes
Keywords: healthy volunteers; antipsychotics; gene expression
MeSH Terms: conditions — Schizophrenia; Diabetes Mellitus | interventions — Olanzapine; ziprasidone

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- olanzapine (Active Comparator): olanzapine
  Interventions: Drug: olanzapine; Drug: ziprasidone
- ziprasidone (Active Comparator): ziprasidone
  Interventions: Drug: olanzapine; Drug: ziprasidone
- Sugar pill (Placebo Comparator): Sugar pill
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: olanzapine — olanzapine 10mg od + placebo od
  Arms: olanzapine; ziprasidone
Drug: ziprasidone — ziprasidone 40mg td
  Arms: olanzapine; ziprasidone
Drug: placebo — placebo td
  Arms: Sugar pill

SUMMARY:
Schizophrenia is a severe chronic and disabling mental disorder and is associated with a significant reduction in life expectancy. Atypical antipsychotic treatment compliance may be jeopardized because of drug induced weight gain and abnormalities in carbohydrate and lipid metabolism.

Aim: to gain data on drug related effects on gene expression and regulation with special regard to glucose metabolism.

ELIGIBILITY:
Inclusion Criteria:

* Male.
* Healthy, defined as absence of relevant diseases.
* Caucasian.
* Aged 18-45 years.
* Body-Mass-Index (BMI): 18-25 kg/m2.
* Signed informed consent.
* No signs of impaired glucose tolerance as evaluated by Oral Glucose Tolerance Test (OGTT) before study inclusion during screening, normal total cholesterol, High Density Lipoprotein (HDL), Low Density Lipoprotein (LDL), triglycerides, normal function of the thyroid. No personal or family history (parents and siblings) of diabetes or other metabolic and relevant diseases as defined by the investigator.
* No indication for psychiatric diseases assessed by structured clinical interview (Mini-International Neuropsychiatric Interview (MINI)).

Exclusion Criteria:

* Personal or family history (parents and siblings) of diabetes or other metabolic diseases, relevant diseases as defined by the investigator.
* History of hypertension, blood pressure > 140/90 at screening, cardiovascular disease.
* Body mass index out of the range of <18 and >25 kg/m.
* Human immunodeficiency virus (HIV) or Hepatitis B/C positive virology.
* Allergy or hypersensitivity against olanzapine/ziprasidone or another excipient.
* Contraindications against the use of the drug according to the Summary of Product Characteristics (SmPC).
* Any drug intake 2 weeks prior to first study day.
* History of excessive bleeding tendency/hemophilia.
* Presence of relevant illness within the last 3 weeks.
* Currently enrolled into an other clinical study with Investigational Medicinal Products (IMPs).
* Last study participation less than 4 weeks.
* Suspected non-compliance with study instructions and life-style requirements.
* History of alcohol or drug abuse.
* Blood/Plasma donation within 4 weeks prior to study day.
* Previous exposure to antipsychotic drugs.
* Nicotine consumption at time of enrolment (at least 3 months of non-smoking required).

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2010-07; Primary Completion 2017-01-01 (Actual); Study Completion 2017-01-01 (Actual)

PRIMARY OUTCOMES:
gene expression profiling | 10 days
  To characterize and compare the gene expression profiles in human subcutaneous adipose and muscle tissue prior and after single dose of olanzapine, ziprasidone and placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Brunner, MD, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Vienna, Austria